CLINICAL TRIAL: NCT05005390
Title: Comparison of Effectiveness of Mask Ventilation and Endotracheal Tube in Pharynx (TTIP) in Patients With Potential Difficult Airway:A Prospective Randomized and Blinded Trial.
Brief Title: Comparison of Effectiveness of Mask Ventilation and Endotracheal Tube in Pharynx (TTIP) in Patients With Potential Difficult Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Travis Markham, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-21-0478
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Results first posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Ventilation Therapy; Complications
Keywords: Bag Mask Ventilation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- TTIP ventilation, then mask ventilation (Experimental): Subjects will first be ventilated with the TTIP technique. If the subjects are adequately ventilated, as defined by carbon dioxide measured during exhalation in at least one of the first three consecutive breaths, ventilation will continue until completion of 10 breaths, for 1 min (Step 1). Subjects will then be ventilated with mask ventilation (Step 2). In Step 1, if ventilation fails with the TTIP technique for all of the first three consecutive breaths, the subject will be crossed over to the mask ventilation. If ventilation fails again with all the first three consecutive breaths after crossover, the study will be terminated. The routine care is resumed including tracheal intubation or laryngeal mask airway (LMA) insertion.
  Interventions: Device: TTIP ventilation; Device: Mask Ventilation
- Mask ventilation, then TTIP ventilation (Active Comparator): Subjects will first be ventilated with the mask technique. If the subjects are adequately ventilated, as defined by carbon dioxide measured during exhalation in at least one of the first three consecutive breaths, ventilation will continue until completion of 10 breaths, for 1 min (Step 1). Subjects will then be ventilated with TTIP technique (Step 2). In Step 1, if ventilation fails for all of the first three consecutive breaths, the subject will be crossed over to the TTIP ventilation. If ventilation fails again with all the first three consecutive breaths after crossover, the study will be terminated. The routine care is resumed including tracheal intubation or LMA insertion.
  Interventions: Device: TTIP ventilation; Device: Mask Ventilation

INTERVENTIONS:
Device: TTIP ventilation — In TTIP ventilation, an endotracheal tube is inserted via the nostril or oral cavity and subsequently advanced until the tip of the tube reaches approximately the level of the glottis.
Device: Mask Ventilation — In mask ventilation, a mask is placed over the nose and mouth.

SUMMARY:
The purpose of this study is to determine the efficacy of TTIP-first ventilation and to compare the efficacy of TTIP first ventilation with the current practice of mask-first ventilation

ELIGIBILITY:
Inclusion Criteria:

* BMI >30 kg/m2
* Mallampati class III or IV
* Requiring general anesthesia

Exclusion Criteria:

* Acute and chronic respiratory disorders, including Chronic obstructive pulmonary disease(COPD)and asthma
* American Society of Anesthesiologists (ASA)physical status classification ≥IV
* Emergency surgery
* Induction requiring rapid sequence for intubation
* Patients requiring awake intubation
* Pregnant women
* Untreated ischemic heart disease
* Contraindication for mask ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Travis Markham, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TTIP Ventilation, Then Mask Ventilation: Subjects will first be ventilated with the TTIP technique. If the subjects are adequately ventilated, as defined by carbon dioxide measured during exhalation in at least one of the first three consecutive breaths, ventilation will continue until completion of 10 breaths, for 1 min (Step 1).Subjects will then be ventilated with mask ventilation (Step 2).In Step 1, if ventilation fails with the TTIP technique for all of the first three consecutive breaths, the subject will be crossed over to the mask ventilation. If ventilation fails again with all the first three consecutive breaths after crossover,the study will be terminated.The routine care is resumed including tracheal intubation or laryngeal mask airway (LMA) insertion.
  TTIP ventilation: In TTIP ventilation, an endotracheal tube is inserted via the nostril or oral cavity and subsequently advanced until the tip of the tube reaches approximately the level of the glottis.
  Mask Ventilation: In mask ventilation, a mask is placed over the nose and mouth.
- Mask Ventilation, Then TTIP Ventilation: Subjects will first be ventilated with the mask technique. If the subjects are adequately ventilated, as defined by carbon dioxide measured during exhalation in at least one of the first three consecutive breaths, ventilation will continue until completion of 10 breaths, for 1 min (Step 1).Subjects will then be ventilated with TTIP technique (Step 2).In Step 1, if ventilation fails for all of the first three consecutive breaths, the subject will be crossed over to the TTIP ventilation. If ventilation fails again with all the first three consecutive breaths after crossover,the study will be terminated.The routine care is resumed including tracheal intubation or LMA insertion.
  TTIP ventilation: In TTIP ventilation, an endotracheal tube is inserted via the nostril or oral cavity and subsequently advanced until the tip of the tube reaches approximately the level of the glottis.
  Mask Ventilation: In mask ventilation, a mask is placed over the nose and mouth.
Period: Overall Study
Arm/Group | TTIP Ventilation, Then Mask Ventilation | Mask Ventilation, Then TTIP Ventilation
Started | 76 | 71
Successfully Completed First Ventilation (Step 1) | 64 | 52
Successfully Completed Second Ventilation (Step 2) | 63 | 63
Completed (Successfully Completed First and Second Ventilation) | 57 | 50
Not Completed | 19 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TTIP Ventilation, Then Mask Ventilation | Mask Ventilation, Then TTIP Ventilation | Total
Number analyzed (Participants) | 76 | 71 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (14.8) | 44.4 (13.0) | 46.2 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 37 | 81
  Male | 32 | 34 | 66
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 76 | 71 | 147
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 36.1 (7.3) | 36.6 (6.0) | 36.3 (6.7)
American Society of Anesthesiology (ASA) Classification [Count of Participants; unit: Participants] — ASA Physical Status Classification System - The purpose of the system is to assess and communicate a patient's pre-anesthesia medical co-morbidities.
  ASA I :A normal healthy patient
  ASA II :A patient with mild systemic disease
  ASA III: A patient with severe systemic disease
  ASA IV: A patient with severe systemic disease that is a constant threat to life
  ASA V: A moribund patient who is not expected to survive without the operation
  ASA VI: A declared brain-dead patient whose organs are being removed for donor purposes
  Participants
    ASA I :A normal healthy patient | 2 | 2 | 4
    ASA II :A patient with mild systemic disease | 31 | 35 | 66
    ASA III: A patient with severe systemic disease | 43 | 33 | 76
    ASA IV: A patient with severe systemic disease that is a constant threat to life | 0 | 1 | 1
    ASA V: A moribund patient who is not expected to survive without the operation | 0 | 0 | 0
    ASA VI: A declared brain-dead patient whose organs are being removed for donor purposes | 0 | 0 | 0
Mallampati Class [Count of Participants; unit: Participants] — The Mallampati class identifies patients at risk for difficult intubation based on the structure of their oropharynx.
  Class I: soft palate, uvula, and pillars are visible
  Class II: soft palate and uvula are visible
  Class III: only the soft palate and base of the uvula are visible
  Class IV: only the hard palate is visible
  Participants
    Class I: soft palate, uvula, and pillars are visible | 24 | 17 | 41
    Class II: soft palate and uvula are visible | 26 | 34 | 60
    Class III: only the soft palate and base of the uvula are visible | 19 | 16 | 35
    Class IV: only the hard palate is visible | 7 | 4 | 11
Provider's training levels [Count of Participants; unit: Participants]
  Attending Anesthesiologists | 9 | 8 | 17
  Anesthesia assistants | 19 | 17 | 36
  Anesthesia residents | 48 | 46 | 94
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  < 30 kg/m^2 | 4 | 3 | 7
  greater than or equal to 30 kg/m^2 to less than 40 kg/m^2(Class 1&2 obesity) | 55 | 54 | 109
  ≥ 40 kg/m^2 (Class 3 obesity) | 17 | 14 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Successful Ventilation
Description: Successful ventilation is defined as expired carbon dioxide with three phases in at least one of the first three consecutive breaths.
Time Frame: from start of ventilation to end of ventilation (about 1 minute)
Population: Data were not collected for 11 participants in the TTIP Ventilation arm and the Mask ventilation arm.
Measure: Count of Participants; unit: Participants
Arm/Group | TTIP Ventilation | Mask Ventilation
Number analyzed (Participants) | 136 | 136
Participants | 127 | 115

2. Secondary Outcome: Expired Tidal Volume of Ventilation
Description: This is measured by readings from the ventilator used in the operating room
Time Frame: from start of ventilation to end of ventilation (about 1 minute)
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | TTIP Ventilation | Mask Ventilation
Number analyzed (Participants) | 107 | 107
ml | 618.22 (313.68) | 719.48 (348.64)

3. Secondary Outcome: Peak Inspiratory Airway Pressure Achieved
Description: This is measured by readings from the ventilator used in the operating room
Time Frame: from start of ventilation to end of ventilation (about 1 minute)
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | TTIP Ventilation | Mask Ventilation
Number analyzed (Participants) | 107 | 107
cmH2O | 19.82 (1.11) | 19.94 (1.76)

4. Secondary Outcome: Dynamic Airway Resistance
Description: This is defined as the peak inspiratory flow divided by the corresponding airway pressure.
Time Frame: from start of ventilation to end of ventilation (about 1 minute)
Population: Data were not collected for this outcome measure.
Arm/Group | TTIP Ventilation | Mask Ventilation
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Satisfaction of the Providers Obtained With Post Ventilation Survey
Time Frame: Baseline before start of surgery
Population: Data were not collected for this outcome measure.
Arm/Group | TTIP Ventilation | Mask Ventilation
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Satisfaction of the Providers Obtained With Post Ventilation Survey
Time Frame: end of surgery (about 1 hour after start)
Population: Data were not collected for this outcome measure.
Arm/Group | TTIP Ventilation | Mask Ventilation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: during time in PACU (about 30 minutes to 2 hours)
Groups:
- TTIP Ventilation: Subjects will first be ventilated with the TTIP technique. If the subjects are adequately ventilated, as defined by carbon dioxide measured during exhalation in at least one of the first three consecutive breaths, ventilation will continue until completion of 10 breaths, for 1 min (Step 1).Subjects will then be ventilated with mask ventilation (Step 2).In Step 1, if ventilation fails with the TTIP technique for all of the first three consecutive breaths, the subject will be crossed over to the mask ventilation. If ventilation fails again with all the first three consecutive breaths after crossover,the study will be terminated.The routine care is resumed including tracheal intubation or laryngeal mask airway (LMA) insertion.
  TTIP ventilation: In TTIP ventilation, an endotracheal tube is inserted via the nostril or oral cavity and subsequently advanced until the tip of the tube reaches approximately the level of the glottis.
  Mask Ventilation: In mask ventilation, a mask is placed over the nose and mouth.
- Mask Ventilation: Subjects will first be ventilated with the mask technique. If the subjects are adequately ventilated, as defined by carbon dioxide measured during exhalation in at least one of the first three consecutive breaths, ventilation will continue until completion of 10 breaths, for 1 min (Step 1).Subjects will then be ventilated with TTIP technique (Step 2).In Step 1, if ventilation fails for all of the first three consecutive breaths, the subject will be crossed over to the TTIP ventilation. If ventilation fails again with all the first three consecutive breaths after crossover,the study will be terminated.The routine care is resumed including tracheal intubation or LMA insertion.
  TTIP ventilation: In TTIP ventilation, an endotracheal tube is inserted via the nostril or oral cavity and subsequently advanced until the tip of the tube reaches approximately the level of the glottis.
  Mask Ventilation: In mask ventilation, a mask is placed over the nose and mouth.
Arm/Group | TTIP Ventilation | Mask Ventilation
All-Cause Mortality (participants affected / at risk) | 0/147 | 0/147
Serious Adverse Events (participants affected / at risk) | 0/147 | 0/147
Other Adverse Events (participants affected / at risk) | 0/147 | 0/147

LIMITATIONS AND CAVEATS:
We calculated the sample size based on a parallel study design that resulted in a sample size of 245. We later performed a sample size calculation based on a crossover study design and realized that by enrolling one hundred forty-seven patients, we would achieve greater than 80% power for our primary analysis to detect a significant difference between the techniques with type I error (α) < 0.05, even with a possible 10% dropout. Therefore, we terminated our study with 147 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT05005390/Prot_SAP_000.pdf